CLINICAL TRIAL: NCT00222196
Title: Oslo Balloon Angioplasty Versus Conservative Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University Hospital, Aker (Other); Pfizer (Industry)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBACT
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-09

CONDITIONS: Peripheral Vascular Disease
Keywords: atherosclerosis; quality of life; pain-score; biomarkers
MeSH Terms: conditions — Peripheral Vascular Diseases; Atherosclerosis

INTERVENTIONS:
Procedure: lifestyle, PTA

SUMMARY:
Background: Percutaneous transluminal angioplasty (PTA) has been popularized as a simple, effective and cheap treatment achieving 50-70% symptomatic patency rates in patients with peripheral occlusive disease.. However, the fact remains that the indication for performing PTA are still more based on opinions than on scientific data.

The purpose of the trial was to randomize patients primarily referred for intermittent claudication into two groups: One group was offered conservative treatment; the other group was offered conservative treatment combined with PTA.

Primary outcome: The patient quality of life. Secondary outcome:Pain-free walking distance; pain-score; death; amputation; changes in relevant biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Age below 75 years
* Symptoms of intermittent claudication with duration > 3 months
* ABPI <0.9
* A two-year follow-up is possible

Exclusion Criteria:

* Subjective pain-free walking distance > 400m
* Critical ischemia
* Previous vascular or endovascular surgery
* Diabetes ulcer
* Other physical disability abrogating organised exercise
* Use of warfarin
* Mentally unable to give informed consent
* Renal insufficiency
* Coagulation disorders Duplex or PTA impossible

Max Age: 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2000-11; Study Completion 2004-12

PRIMARY OUTCOMES:
The patient quality of life.

SECONDARY OUTCOMES:
Pain-free walking distance; pain-score; death; amputation; changes in relevant biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Marthe Nylaende, MD, Principal Investigator — Aker and Ullevål University Hospitals, Oslo, Norway